CLINICAL TRIAL: NCT04490148
Title: Remote Pulmonary Function Testing and Nurse Respiratory Health Coaching in Amyotrophic Lateral Sclerosis
Brief Title: Remote Pulmonary Function Testing and Nurse Coaching in ALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: ALS Association (Other)
Responsible Party: Principal Investigator, Zachary Simmons, MD, Professor of Neurology and Humanities, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00006924part2
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: ALS
Keywords: Telemedicine; Pulmonary Function Testing; Telehealth

STUDY DESIGN:
Intervention Model Description: A longitudinal parallel group study of repeated measures of remote PFTs, nurse coaching, and their impact on respiratory outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- remote PFT (rPFT) longitudinal (Active Comparator): Subjects will undergo standard pulmonary function testing as part of standard clinical procedure. They will also undergo weekly remote pulmonary function testing using the telemedicine interface and study equipment.
  Interventions: Device: remote pulmonary function testing; Device: standard pulmonary function testing
- remote PFT (rPFT) + Nurse Coaching longitudinal (Experimental): Subjects will undergo standard pulmonary function testing as part of standard clinical procedure. They will also undergo weekly remote pulmonary function testing using the telemedicine interface and study equipment, and receive monthly coaching from an ALS nurse.
  Interventions: Device: remote pulmonary function testing; Device: standard pulmonary function testing; Behavioral: Nurse Respiratory Health Coaching (NRHC)

INTERVENTIONS:
Device: remote pulmonary function testing — Telemedicine delivery of pulmonary function testing in ALS, including Forced Vital Capacity (FVC) and Maximal Inspiratory Pressure (MIP)
Device: standard pulmonary function testing — Standard clinical delivery of pulmonary function testing in ALS, including Forced Vital Capacity (FVC) and Maximal Inspiratory Pressure (MIP)
Behavioral: Nurse Respiratory Health Coaching (NRHC) — Nurse Respiratory Health Coaching - The NRHC intervention follows the "teamlet" model described by Bennett et al. [Bennett2010], made up of the research coordinator who performs respiratory testing, and the nurse practitioner who coaches using the GROW (goals, realities, options, wrap-up) model.
  Arms: remote PFT (rPFT) + Nurse Coaching longitudinal

SUMMARY:
Comparison of respiratory outcomes in patients receiving telemedicine-guided remote pulmonary function testing (rPFT) with or without the additional support of nurse coaching. This is a randomized controlled study which assesses the effects rPFT and coaching on respiratory outcomes and quality of life.

DETAILED DESCRIPTION:
This is a two-arm, randomized study to determine 1) whether weekly monitoring of respiratory function can lead to timelier initiation of NIV and 2) whether structured nurse coaching leads to improved self-efficacy for managing disease and better maintenance of respiratory health. For enrollees in both arms, standard FVC and MIP measurements obtained approximately every three months by the respiratory therapist during ALS Clinic are supplemented with self-administered rPFTs performed weekly. Enrollees in the rPFT+NRHC (nurse respiratory health coaching) arm will additionally receive monthly coaching with the study nurse via telehealth. Outcomes include measures of quality of life and self-efficacy for managing disease.

ELIGIBILITY:
Inclusion Criteria:

Patients:

1. Possess a diagnosis of definite, probable, probable laboratory-supported, or possible ALS by revised El Escorial research criteria [Brooks2000].
2. Be 18 years of age or older.
3. Have a caregiver available to participate in the study
4. Symptom onset within the last three years.
5. Have a computer and home internet service sufficient for engaging in telemedicine sessions.
6. Have a second device capable of downloading the spirometer application from an app store (Android- or iOS-based smartphone or tablet).

Caregivers:

1. Be 18 years of age or older, of either gender.
2. Be able and willing to provide informed consent.

Exclusion Criteria:

Patients:

1. Use of NIV or diaphragm pacer at time of obtaining informed consent.
2. FVC ≤50% predicted or MIP > -60 cm of water.
3. ALS Functional Rating Scale (ALSFRS-R) [Cedarbaum1999] score on day of screening of ≥2 on items for speech, swallowing, and salivation. These items are indicators of bulbar dysfunction, which limits the reliability of PFT administration.
4. Cognitive impairment, as judged by the ALS clinic neurologist, that prevents participation in the study.

Caregivers: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hershey Medical Center ALS Clinic, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plan at this time to share data with other researchers

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 5 participants exited the study prior to randomization.
Groups:
- Remote Pulmonary Function Testing (rPFT) Longitudinal: Subjects will undergo standard pulmonary function testing as part of standard clinical procedure. They will also undergo weekly remote pulmonary function testing using the telemedicine interface and study equipment.
  remote pulmonary function testing: Telemedicine delivery of pulmonary function testing in ALS, including Forced Vital Capacity (FVC) and Maximal Inspiratory Pressure (MIP)
  standard pulmonary function testing: Standard clinical delivery of pulmonary function testing in ALS, including Forced Vital Capacity (FVC) and Maximal Inspiratory Pressure (MIP)
- Remote Pulmonary Function Testing (rPFT) + Nurse Coaching Longitudinal: Subjects will undergo standard pulmonary function testing as part of standard clinical procedure. They will also undergo weekly remote pulmonary function testing using the telemedicine interface and study equipment, and receive monthly coaching from an amyotrophic lateral sclerosis (ALS) nurse.
  remote pulmonary function testing: Telemedicine delivery of pulmonary function testing in ALS, including Forced Vital Capacity (FVC) and Maximal Inspiratory Pressure (MIP)
  standard pulmonary function testing: Standard clinical delivery of pulmonary function testing in ALS, including Forced Vital Capacity (FVC) and Maximal Inspiratory Pressure (MIP)
  Nurse Respiratory Health Coaching (NRHC): Nurse Respiratory Health Coaching - The NRHC intervention follows the "teamlet" model described by Bennett et al. [Bennett2010], made up of the research coordinator who performs respiratory testing, and the nurse practitioner who coaches using the GROW (goals, realities, options, wrap-up) model.
Period: Overall Study
Arm/Group | Remote Pulmonary Function Testing (rPFT) Longitudinal | Remote Pulmonary Function Testing (rPFT) + Nurse Coaching Longitudinal
Started | 12 | 17
Completed | 11 | 12
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Remote PFT (rPFT) Longitudinal | Remote PFT (rPFT) + Nurse Coaching Longitudinal | Total
Number analyzed (Participants) | 12 | 17 | 29
Age, Continuous [Median (Full Range); unit: years] | 61 [45 to 69] | 65 [55 to 79] | 64 [45 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 14
  Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 17 | 29

OUTCOME MEASURES:

1. Primary Outcome: Date of Identification of Noninvasive Ventilation (NIV) Need From rPFT Monitoring
Description: NIV is typically prescribed when an individual demonstrates signs of respiratory failure. In this study, forced vital capacity (FVC) of 50% or less of the predicted value serves as a surrogate for respiratory failure and constitutes identification of NIV need. First date of remote measurement of FVC 50% or less of the predicted value is reported here.
Time Frame: 1 year
Population: Subset of patients include those who have a date of identification of NIV need from both remote PFT monitoring and standard PFT monitoring. Groups are combined because inferences across groups with respect to this outcome were not planned and are not reported.
Measure: Median (Full Range); unit: days after enrollment
Groups:
- Total Group: The full cohort from both arms of the study. There was no comparison of the primary outcome across groups.
Arm/Group | Total Group
Number analyzed (Participants) | 7
days after enrollment | 176 [36 to 365]

2. Primary Outcome: Date of Identification of NIV Need From Standard PFT Monitoring
Description: NIV is typically prescribed when an individual demonstrates signs of respiratory failure. In this study, forced vital capacity (FVC) of 50% or less of the predicted value serves as a surrogate for respiratory failure and constitutes identification of NIV need. First date of standard, in-clinic measurement of FVC 50% or less of the predicted value is reported here.
Time Frame: From date of enrollment until first identification of non-invasive ventilation need, assessed up to 1.5 years
Population: Subset of patients include those who have a date of identification of NIV need from both remote PFT monitoring and standard monitoring.
Measure: Median (Full Range); unit: days after enrollment
Groups:
- Total Group: Total of participants in both arms of the study
Arm/Group | Total Group
Number analyzed (Participants) | 7
days after enrollment | 259 [76 to 413]

3. Primary Outcome: Self-efficacy for Managing Medications and Treatments
Description: The self-efﬁcacy assessment contains questions from the Patient-Reported Outcomes Measurement Information System (PROMIS) item banks on Self-Efficacy for Managing Medications and Treatments (4 items). Cumulative T-scores from each test bank were reported at months 0, 3, 6, 9, and 12, with a mean score of 50±10, higher numbers indicating greater self-efficacy. The reported value is the slope of regression of self-efficacy on time, in T-score points per month.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: points per month
Arm/Group | Remote PFT (rPFT) Longitudinal | Remote PFT (rPFT) + Nurse Coaching Longitudinal
Number analyzed (Participants) | 12 | 17
points per month | -.238 (.393) | .474 (1.583)

4. Primary Outcome: Self-efficacy for Managing Social Interactions
Description: The self-efﬁcacy assessment contains questions from the PROMIS item bank on Self-Efficacy for Managing Social Interactions (5 items). Cumulative T-scores from each test bank were reported at months 0, 3, 6, 9, and 12, with a mean score of 50±10, higher numbers indicating greater self-efficacy. The reported value is the slope of regression of self-efficacy on time, in T-score points per month.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: points per month
Arm/Group | Remote PFT (rPFT) Longitudinal | Remote PFT (rPFT) + Nurse Coaching Longitudinal
Number analyzed (Participants) | 12 | 17
points per month | -.041 (.551) | -.181 (.688)

5. Primary Outcome: Self-efficacy for Managing Symptoms
Description: The self-efﬁcacy assessment contains questions from the PROMIS item bank on Self-Efﬁcacy for Managing Symptoms (9 items). Cumulative T-scores from each test bank were reported at months 0, 3, 6, 9, and 12, with a mean score of 50±10, higher numbers indicating greater self-efficacy. The reported value is the slope of regression of self-efficacy on time, in T-score points per month.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: points per month
Arm/Group | Remote PFT (rPFT) Longitudinal | Remote PFT (rPFT) + Nurse Coaching Longitudinal
Number analyzed (Participants) | 12 | 17
points per month | -.279 (.636) | -.255 (.813)

6. Secondary Outcome: Dyspnea Characteristics
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Pool v1.0 - Dyspnea Characteristics (5 items), which uses Likert-type scaling that are summed to a total score. Participants complete this questionnaire each month (12 total administrations). Total score range 0-44, with higher numbers indicating more severe dyspnea. The reported value is the slope of regression of total score on time, in point change per month.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: points per month
Arm/Group | Remote Pulmonary Function Testing (rPFT) Longitudinal | Remote Pulmonary Function Testing (rPFT) + Nurse Coaching Longitudinal
Number analyzed (Participants) | 12 | 17
points per month | .029 (.408) | .272 (.964)

7. Secondary Outcome: Respiratory-related Symptoms
Description: Subjects were asked to report whether they experienced the following symptoms in the past month during each month on the study (12 administrations): excessive secretions, drooling, choking on secretions, morning headache. Reported value is the sum of experienced symptoms (0-4) summed over 12 months. Participants could experience none of these symptoms (0) up to experiencing all symptoms each month (48).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: number of symptoms reported
Arm/Group | Remote Pulmonary Function Testing (rPFT) Longitudinal | Remote Pulmonary Function Testing (rPFT) + Nurse Coaching Longitudinal
Number analyzed (Participants) | 12 | 17
number of symptoms reported | 11.4 (6.4) | 7.6 (6.0)

8. Secondary Outcome: rPFT Adherence
Description: Participant adherence to rPFT protocol, defined as the percentage of eligible weeks with a submitted rPFT report.
Time Frame: 1 year
Measure: Median (Full Range); unit: Percentage
Groups:
- Total Group: The full cohort from both arms of the study. There was no comparison performed across groups for this outcome.
Arm/Group | Total Group
Number analyzed (Participants) | 29
Percentage | 82.2 [36.7 to 99.0]

9. Secondary Outcome: Dyspnea Functional Limitations
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v1.0 - Dyspnea Functional Limitations - Short Form 10a (10 items), which uses Likert-type scaling that are summed to a total score. Participants complete this questionnaire each month (12 total administrations). Total score range 0-30, with higher numbers indicating more functional limitations due to dyspnea. The reported value is the slope of regression of total score on time, in point change per month.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: points per month
Arm/Group | Remote Pulmonary Function Testing (rPFT) Longitudinal | Remote Pulmonary Function Testing (rPFT) + Nurse Coaching Longitudinal
Number analyzed (Participants) | 12 | 17
points per month | -.022 (.350) | -.255 (.838)

10. Secondary Outcome: Sleep Related Impairment
Description: Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank v1.0 - Sleep Related Impairment - Short Form 8a (8 items), which uses Likert-type scaling that are summed to a total score. Participants complete this questionnaire each month (12 total administrations). Total score range 8-40, with higher numbers indicating more sleep-related impairment. The reported value is the slope of regression of total score on time, in point change per month.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: points per month
Arm/Group | Remote Pulmonary Function Testing (rPFT) Longitudinal | Remote Pulmonary Function Testing (rPFT) + Nurse Coaching Longitudinal
Number analyzed (Participants) | 12 | 17
points per month | .095 (.320) | .140 (.523)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at site visits as well as through participant self report between visits while the subject was on the study. This occurred over the course of one year on average.
Arm/Group | Remote PFT (rPFT) Longitudinal | Remote PFT (rPFT) + Nurse Coaching Longitudinal
All-Cause Mortality (participants affected / at risk) | 1/12 | 2/17
Serious Adverse Events (participants affected / at risk) | 1/12 | 6/17
Other Adverse Events (participants affected / at risk) | 0/12 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Remote PFT (rPFT) Longitudinal (N=12) | Remote PFT (rPFT) + Nurse Coaching Longitudinal (N=17)
Death due to respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anasarca (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fall and Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT04490148/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT04490148/ICF_001.pdf